CLINICAL TRIAL: NCT01865123
Title: A Randomized Controlled Trial of Meditation Compared to Exposure Therapy and Education Control on PTSD in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency); Maharishi University of Management Research Institute (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sanford Nidich, Ed.D., Associate Director, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT110413
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; transcendental meditation; cognitive behavioral therapy; prolonged exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Meditation; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transcendental Meditation (Experimental): TM is a simple, natural, effortless mental technique practiced with eyes closed sitting for 20 minutes twice a day. This allows the practitioner to experience lesser excited levels of the mind and correspondingly greater degrees of physical relaxation. TM is a traditional meditation technique that has its origin in the ancient Vedic tradition of India.
  Interventions: Behavioral: Transcendental Meditation
- Prolonged Exposure (Active Comparator): Prolonged Exposure (PE) is a specialized type of Cognitive Behavorial Therapy employing a manualized, trauma-focused behavioral treatment for PTSD and is based on exposure principles and emotional processing theory.
  Interventions: Behavioral: Prolonged Exposure
- Educational Control (Placebo Comparator): Didactic based instructional classes will provide health education which will include the benefits of proper diet, exercise, and reducing smoking and alcohol. No stress management techniques will be taught.
  Interventions: Behavioral: Educational control

INTERVENTIONS:
Behavioral: Transcendental Meditation — A standard 7 step course will be offered including an introductory and preparatory lectures, personal one-on-one instruction with a certified TM teacher followed by 3 consecutive days of classes on how to meditate correctly and effortlessly, how to understand mechanisms of stress release and sequential development to higher levels of human consciousness and enjoying ones full potential. Followup meetings will provide checking of TM practice, sharing of group experiences with the TM practice and knowledge to motivate and inspire continued regularity with the practice. The certified TM instructor will have experience with PTSD in this veteran population.
  Other Names: meditation, mantra meditation, stress management
  Arms: Transcendental Meditation
Behavioral: Prolonged Exposure — Prolonged exposure therapy, a specific form of cognitive behavioral therapy, is considered the standard psychotherapy treatment for PTSD . The delivery of PE will be by a trained study therapist. There will be 16 individual sessions provided to each participant. Homework will include relaxation and breathing exercises and anxiety diaries.
  Other Names: Cognitive Behavioral Therapy
  Arms: Prolonged Exposure
Behavioral: Educational control — This group will receive group-administered didactic health education specific to the PTSD veterans population. It will include emphasis on healthy lifestyle changes to promote more positive mental and physical health. The classes will be matched with the TM and PE interventions to control for time, instructor attention and other non-specific factors.
  Other Names: Health Education
  Arms: Educational Control

SUMMARY:
The purpose of this study is to compare the effectiveness of the Transcendental Meditation (TM) program to the more standard Cognitive Behavioral Therapy with Prolonged Exposure (CBT-PE) in treating posttraumatic stress disorder (PTSD) in war Veterans over a three month treatment period.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a common and debilitating anxiety condition that affects up to 20% of war Veterans. PTSD is often a chronic problem for Veterans, affecting reintegration into society, family and marital relationships, sleep, employment stability, substance abuse rates, and risk for depression and suicide, among other areas. Although several effective therapies exist to treat PTSD, research shows that up to half of patients completing these treatments continue to have elevated symptoms indicating the important need for developing additional treatment options.

In the current trial, we propose to test one such new treatment, specifically a meditation practice known as Transcendental Meditation. The Transcendental Meditation (TM) program will be compared to one of the best and most standard of PTSD therapies (Prolonged Exposure therapy), and a educational control group. This study will recruit 210 War Veterans clinically diagnosed with PTSD from the San Diego VA Healthcare System over a 4 year study period.

The intervention period will be 3 months. Study participants will be randomized equally to one of three study groups, either

1. Transcendental Meditation (TM) or
2. Cognitive Behavioral Therapy with Prolonged Exposure (CBT-PE) or
3. Educational control group.

The primary outcome will be scores on the Clinically Administered PTSD Scale (CAPS).

Secondary outcomes will includes scores on PTSD symptoms including depression, anger, mood disturbance and quality of life.

Behavioral or lifestyle factors will also be measured including smoking, alcohol, and non-described drug usage along with compliance with each treatment.

Physiological markers of stress and disease risk will include cortisol, blood pressure, inflammatory markers and body mass.

If successful, these research findings will serve to provide key data on the feasibility and efficacy of the TM program as an alternative therapy for PTSD. The results will serve to inform policy decisions on the study and application of standardized and validated stress reduction programs in veteran populations.

ELIGIBILITY:
Inclusion Criteria:

1. Current medical diagnosis of PTSD
2. A symptom severity score of 45 or higher on the Clinically Administered PTSD Scale (CAPS)
3. Three or more months since service-related trauma
4. If being treated with psychoactive medication, a stable regimen (no change in drugs or dose) for at least 2 months before enrollment
5. Age: 18 years or older
6. Language: English literate -

Exclusion Criteria:

1. Current unstable or uncontrolled psychotic symptoms, mania or bipolar disorder 2. Current suicidal or homicidal ideation 3. Moderate or greater cognitive impairment indicated by chart diagnosis or observable cognitive difficulties 4. Having received Prolonged Exposure therapy or having been instructed in Transcendental Meditation.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Clinically Administered PTSD Scale (CAPS) | 3 months
  This scale is currently the gold standard for assessing the severity of post-traumatic stress disorder (PTSD) using a face-to-face interview with the patient and a professionally trained medical/psychiatric administrator.

SECONDARY OUTCOMES:
Self-Report Symptoms of PTSD | 3 months
  The PTSD Checklist- Military version (PCL-M) will assess PTSD symptoms in response to stressful military experiences.
  The Patient Health Questionnaire (PHQ)-9 will be used to evaluate clinical depression.
  The Profile of Mood States (POMS - will be used to evaluate total mood disturbance (TMD) main scale and tension/anxiety, depression/dejection, and anger/hostility subscales.
  The Social Support Questionnaire (SSQ) will be used to evaluate level of social support.
  The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form will used to assess overall quality of life.

OTHER OUTCOMES:
Behavioral Measures | 3 months
  For substance usage, participants will be evaluated by the Weekly Recall (WR) method on alcohol, non-prescribed drugs, and smoking
Biomarkers of Stress | 3 months
  Blood Pressure will be measured three times with a mercury sphygmomanometer after five minutes rest. Three readings will be taken one minute apart. The latter two will be averaged for clinic visit mean.
  Participants will complete a 24-hour urine collection for catecholamine levels as a marker of chronic sympathetic nervous system activation and cortisol as a marker for hypothalamic-pituitary-adrenal (HPA) axis activation.
  Inflammatory biomarkers relevant to PTSD and cardiovascular disease will be assayed including C-Reactive Protein(CRP), Tumor Necrosis Factor(TNF-a), and Interleukin-6(IL-6).
Treatment Adherence | 3 months
  Adherence with the study interventions will be assessed through multiple measures in the two study groups. Adherence with health education and the stress reduction practice will be measured by: 1) daily home practice logs; 2) basic and follow-up meetings attended; and 3) random phone calls to participants by staff to determine recent practice of participants' respective programs. The Patient Satisfaction Questionnaire will also be used to evaluate the TM and CBT-PE programs.

CONTACTS AND LOCATIONS:
Overall Officials: Sanford I Nidich, EdD, Principal Investigator — Maharishi University of Management Research Institute; Thomas Rutledge, PhD, Principal Investigator — San Diego VA Healthcare System
Locations (1):
- San Diego VA Healthcare System, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rutledge T, Nidich S, Schneider RH, Mills PJ, Salerno J, Heppner P, Gomez MA, Gaylord-King C, Rainforth M. Design and rationale of a comparative effectiveness trial evaluating transcendental meditation against established therapies for PTSD. Contemp Clin Trials. 2014 Sep;39(1):50-6. doi: 10.1016/j.cct.2014.07.005. Epub 2014 Jul 25. PMID 25066921
- [Result] Nidich S, Mills PJ, Rainforth M, Heppner P, Schneider RH, Rosenthal NE, Salerno J, Gaylord-King C, Rutledge T. Non-trauma-focused meditation versus exposure therapy in veterans with post-traumatic stress disorder: a randomised controlled trial. Lancet Psychiatry. 2018 Dec;5(12):975-986. doi: 10.1016/S2215-0366(18)30384-5. Epub 2018 Nov 15. PMID 30449712